CLINICAL TRIAL: NCT06796426
Title: A Treatment Protocol for the Use of Plozasiran in Adults With Familial Chylomicronemia Syndrome (FCS). A Single Patient Protocol for the Use of Plozasiran In Adolescents With Familial Chylomicronemia Syndrome (FCS).
Brief Title: Treatment Protocol of Plozasiran in Adults and Adolescents With FCS
Status: Available | Type: Expanded Access
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: AROAPOC3-EAP-002; AROAPOC3-EAP-003 (Other: Arrowhead Pharmaceuticals Inc)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Familial Chylomicronemia
MeSH Terms: conditions — Hyperlipoproteinemia Type I | interventions — plozasiran

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Plozasiran — 25 mg ARO-APOC3 by sc injection administered by healthcare professional
  Other Names: ARO-APOC3

SUMMARY:
This is a treatment program for the use of plozasiran in adults (AROAPOC3-EAP-002) and adolescents (AROAPOC3-EAP-003) with familial chylomicronemia syndrome (FCS). The program will enroll eligible patients ≥15 years of age, with fasting triglycerides ≥880 mg/dL (≥10 mmol/L) that is not adequately controlled with standard lipid-lowering therapy, and with a diagnosis of FCS. Patients will receive 25 mg of plozasiran by subcutaneous (sc) injection on Day 1 and every three months for a total of 5 injections. The duration of the program is 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Fasting triglycerides (TG) ≥ 880mg/dL that is not sufficiently controlled on standard lipid-lowering therapy
* Established diagnosis of FCS based on documented history of fasting TG levels in excess of 1000 mg/dL on repeated testing (for at least 3 prior occasions), and at least one of the following: a supportive genetic test, documented history of recurrent episodes of acute pancreatitis not caused by alcohol or cholelithiasis, documented history of recurrent hospitalizations for severe abdominal pain without other explainable cause, documented history of childhood pancreatitis, family history of hypertriglyceridemia-induced pancreatitis
* Willing to follow dietary counseling based on local standard of care, consistent with an intake of ≤ 20 g of fat per day
* If on medications for management of type 2 diabetes the dosing regimen must be stable.
* Participants of childbearing potential must agree to use a highly effective form of contraception in addition to a male condom during the program and for at least 90 days after the last dose of plozasiran

Exclusion Criteria:

* Diabetes mellitus with any of the following at Day 1: newly diagnosed within the past 24 weeks, HbA1c ≥9.0% within the past 4 weeks, meaningful medical events relating to poor glycemic control, changes in basal insulin regimen of more than =/- 10 units within 12 weeks if insulin-dependent
* Clinical evidence of primary hypothyroidism, primary subclinical hypothyroidism, or secondary hypothyroidism
* History of bleeding diathesis or coagulopathy
* Current diagnosis of nephrotic syndrome
* Eligible to receive any commercially available FDA-approved therapeutic for treatment of FCS unless proven to be ineffective or judged inappropriate by the treating physician
* History of acute coronary syndrome events (adults with FCS only)
* New York Heart Association Class III or IV heart failure or last known ejection fraction of <30% (adults with FCS only)
* History of stroke, transient ischemic attack, or peripheral artery disease within 24 weeks of first dose (adults with FCS only) Note: Additional inclusion/exclusion criteria may apply per protocol

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Arrowhead Pharmaceuticals, Inc., Pasadena, California, United States

REFERENCES:
- See also: Related Info — https://arrowheadpharma.com/patients-caregivers/expanded-access-programs/